CLINICAL TRIAL: NCT04781855
Title: Ipilimumab Combined With Ibrutinib and Nivolumab for Patients With Chronic Lymphocytic Leukemia (CLL) and Richter Transformation (RT)
Brief Title: Ipilimumab, Ibrutinib, and Nivolumab for the Treatment of Chronic Lymphocytic Leukemia and Richter Transformation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0% Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0571; NCI-2020-14161 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0571 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Richter Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (ipilimumab, ibrutinib) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 1 of cycle 1, patients also receive ibrutinib PO QD in the absence of disease progression or unacceptable toxicity. Patients who complete 4 doses of ipilimumab and are deriving benefit from it, without severe toxicities, may continue to receive ipilimumab every 12 weeks for up to a total of 2 years.
  Interventions: Drug: Ibrutinib; Biological: Ipilimumab
- Part B (ipilimumab, nivolumab, ibrutinib) (Experimental): Patients receive ipilimumab IV over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 7 of cycle 1, patients also receive ibrutinib PO QD in the absence of disease progression or unacceptable toxicity. Patients who complete 4 doses of ipilimumab and nivolumab, and are deriving benefit from it, without severe toxicities, may continue to receive ipilimumab every 12 weeks and nivolumab every 4 weeks for up to a total of 2 years.
  Interventions: Drug: Ibrutinib; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Part B (ipilimumab, nivolumab, ibrutinib)

SUMMARY:
This phase I/Ib trial evaluates the best dose and side effects of ipilimumab in combination with either ibrutinib alone or with ibrutinib and nivolumab in treating patients with chronic lymphocytic leukemia (CLL) and Richter transformation (RT). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving ipilimumab with either ibrutinib alone or with ibrutinib and nivolumab may help control CLL and RT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of ipilimumab in combination with ibrutinib in patients with CLL/small lymphocytic lymphoma (SLL)/RT. (Part A) II. To determine the MTD and DLT of ipilimumab in combination with nivolumab and ibrutinib in patients with CLL/SLL/RT. (Part B)

SECONDARY OBJECTIVES:

I. To determine the efficacy (response rate, defined as complete response [CR] + complete response with incomplete marrow recovery [CRi] + partial response [PR]) of the combination therapy.

II. To determine the progression-free survival and overall survival of the combination therapy.

EXPLORATORY OBJECTIVE:

I. To study immunological and molecular changes in peripheral blood, lymph node, and bone marrow in response to the combination therapy.

OUTLINE: This is a dose-escalation study of ipilimumab followed by a dose-expansion study. Patients are assigned to 1 of 2 parts.

PART A: Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 1 of cycle 1, patients also receive ibrutinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity. Patients who complete 4 doses of ipilimumab and are deriving benefit from it, without severe toxicities, may continue to receive ipilimumab every 12 weeks for up to a total of 2 years.

PART B: Patients receive ipilimumab IV over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 7 of cycle 1, patients also receive ibrutinib PO QD in the absence of disease progression or unacceptable toxicity. Patients who complete 4 doses of ipilimumab and nivolumab, and are deriving benefit from it, without severe toxicities, may continue to receive ipilimumab every 12 weeks and nivolumab every 4 weeks for up to a total of 2 years.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Patients with a diagnosis of CLL or SLL, refractory to and/or relapsed after at least one prior therapy (prior therapy could be a chemoimmunotherapy regimen, or a targeted therapy such as a BTK inhibitor, a BCL2 inhibitor, or a PI3 kinase inhibitor) or untreated with del(17p) by fluorescence in situ hybridization (FISH) (high-risk cytogenetics) and have an indication for treatment by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria
* Cohort 2: Patients with a diagnosis of CLL or SLL who have been on ibrutinib for at least 9 months with measurable persistent disease (absolute lymphocyte count [ALC] > 4K/uL, any lymph node > 1.5 cm by computed tomography [CT] scan, or > 30% lymphocytes on bone marrow aspirate differential)
* Cohort 3: Patients with a diagnosis of RT
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x upper limit of normal (ULN). For patients with Gilbert's disease, total bilirubin up to =< 3 x ULN is allowed provided normal direct bilirubin
* Serum creatinine =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (unless deemed to be disease related)
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-human chorionic gonadotropin [hCG]) pregnancy test result within 14 days prior to the first dose of treatment and must agree to use an effective contraception method during the study and for 23 weeks following the last dose of the study drugs. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drugs
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses). If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center and after consultation with the principal investigator
* Any major surgery, radiotherapy, cytotoxic chemotherapy, biologic therapy, immunotherapy, immunomodulatory drugs, experimental therapy within 4 weeks prior to the first dose of the study drugs. Note: Prior therapy with anti CD20 monoclonal antibody, anti CD52 monoclonal antibody, and lenalidomide are allowed. For oral targeted therapies (such as idelalisib, venetoclax), a washout of 3 days is allowed. For patients who are on ibrutinib at study entry - may continue ibrutinib without interruption
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 2 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional classification
* History of stroke or cerebral hemorrhage within 2 month
* Patients who have uncontrolled hypertension (defined as sustained systolic blood pressure >= 140 mmHg or diastolic >= 90 mmHg)
* Known evidence of active cerebral/meningeal CLL. Patients may have history of central nervous system (CNS) leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of registration
* Active, uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring steroid therapy
* Patients with autoimmune diseases are excluded: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus, Wegener's granulomatosis)
* Patients with previous allogeneic stem cell transplant (SCT) within 6 months or with active acute or chronic graft-versus host disease are excluded. Patients must be off immunosuppression for graft versus host disease (GVHD) for at least 30 days before cycle 1 day 1
* Patients with organ allografts (such as renal transplant) are excluded
* History of interstitial lung disease or pneumonitis
* Patients who are on high dose steroids (> 10 mg daily of prednisone or equivalent) or immune suppression medications. Note: Patients on high-dose steroids (doses > 10 mg/day of prednisone or equivalent) or immune suppression medications are eligible provided these drugs are discontinued at least 3 days prior to starting on the study drugs
* Patients with uncontrolled active infection (viral, bacterial, and fungal) are not eligible
* Current or chronic hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Patient is pregnant or breast-feeding
* Concurrent use of investigational therapeutic agent
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ipilimumab | Up to 2 years
Dose limiting toxicities | During first 21 days on study intervention
  DLT is defined as clinically significant non-hematologic adverse event or abnormal laboratory value assessed as unrelated to disease, intercurrent illness, or concomitant medications and occurring during the first 21 days.

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years
  Defined as complete response (CR) + complete response with incomplete marrow recovery (CRi) + partial response (PR). Response will be assessed by the investigator, based on physical examinations, computed tomography scans, laboratory results, and bone marrow examinations, according to the modified 2008 International Workshop on Chronic Lymphocytic Leukemia response criteria for chronic lymphocytic leukemia. The overall response rate (i.e., CR/CRi/PR) will be estimated along with the exact 95% confidence interval.
Progression-free survival | From treatment start date until the date of disease progression date or death due to any cause, whichever occurred first, assessed up to 2 years
  Assessed using Kaplan-Meier method.
Overall survival | From treatment start date until the date of death due to any cause, assessed up to 2 years
  Assessed using Kaplan-Meier method.
Incidence of adverse events | Up to 2 years
  Will be summarized by treatment, category, severity and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04781855/ICF_000.pdf